CLINICAL TRIAL: NCT02907944
Title: Working With HIV Clinics to Adopt Addiction Treatments Using Implementation Facilitation (WHAT-IF?)
Brief Title: Working With HIV Clinics to Adopt Addiction Treatments Using Implementation Facilitation
Acronym: WHAT-IF?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HIC1509016500; R01DA041067 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Substance-related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care- Control (No Intervention): We will use a stepped wedge design to evaluate the effect of the Implementation Facilitation on the outcomes. The first phase for all clinics is a control phase where clinic staff and patients engage in usual care. The time to implementation is randomly assigned. Each clinic is then followed prospectively to determine their outcome status.
- Implementation Facilitation (Experimental): We will use a stepped wedge design to evaluate the effect of the Implementation Facilitation on the outcomes. The time to implementation in a stepped wedge design is randomly assigned. Clinics are then followed prospectively to determine their outcome status..
  Interventions: Behavioral: Implementation Facilitation

INTERVENTIONS:
Behavioral: Implementation Facilitation — Implementation Facilitation is an evidence-based strategy tailored to the specific needs of the clinic, designed to increase uptake of evidence based treatments for tobacco, alcohol and opioid use disorders. Will include provider education and academic detailing.
  * External Facilitator: Outside content expert who assists site
  * Local Champion: Site stakeholder who promotes change
  * Provider Education and Academic Detailing: Provision of unbiased peer education
  * Stakeholder Engagement: Aligning goals of implementation and those impacted
  * Tailor Program to Site: Addressing site specific needs based on Aim 1
  * Performance Monitoring and Feedback: Assess implementation of screening and treatment efforts and inform site of results
  * Formative Evaluation: Quant. and qual. determination of impact
  * Establish a Learning Collaborative: Shared learning opportunities tailored to stakeholders
  * Program Marketing: Increase attention to availability of on-site addiction treatment services
  Arms: Implementation Facilitation

SUMMARY:
Tobacco, alcohol and opioid use disorders threaten the health of HIV-infected patients. What if evidence-based counseling and medication treatments for tobacco, alcohol and opioid use disorders (herein refered to as addiction treatments) were routinely provided in HIV clinics? Implementation Facilitation is an established strategy to increase the uptake of evidence-based treatments. Our goal is to evaluate the impact of Implementation Facilitation on the use of addiction treatments in four large HIV clinics.

The purpose of the WHAT-IF study is:

Aim 1. Among key stakeholders, to use quantitative and qualitative (mixed) methods to identify the site-specific evidence, context and facilitation-related barriers and facilitators to the integration of addiction treatments to help tailor an Implementation Facilitation for each clinic.

Aim 2. To evaluate the impact of Implementation Facilitation on:

2a: Organizational readiness to deliver addiction treatments 2b: Provider readiness to deliver addiction treatments 2c: Provision of addiction treatments 2d: Changes in organizational models of care used to deliver addiction treatments

Aim 3. To evaluate the impact of Implementation Facilitation on antiretroviral therapy receipt, HIV viral suppression, VACS Index, and retention in HIV care among patients eligible for addiction treatment.

DETAILED DESCRIPTION:
The Working with HIV clinics to adopt Addiction Treatments using Implementation Facilitation (WHAT IF?) study will evaluate the impact of Implementation Facilitation on the adoption of addiction treatment services in four HIV clinics. We will use a stepped wedge design . The primary comparison is of the change that occurs from the pre-implementation period to two post-implementation periods, the initial six months (evaluation) and the following six months (maintenance). This proposal will consist of three main components in each of four clinics: 1) formative evaluation with key stakeholders at each site to guide and refine the Implementation Facilitation, 2) conduct of the Implementation Facilitation and 3) an evaluation of the impact of the Implementation Facilitation on organization and provider-level readiness, provision of addiction treatments, and HIV outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria:

* HIV-infected
* Receiving HIV care in the index clinic
* Age >18 years old
* Meets criteria for lifetime or current tobacco, alcohol and/or opioid use disorder regardless of addiction treatment status
* Able to provide verbal informed consent

Staff inclusion criteria:

* Employed at participating HIV clinic for at least 6 months
* Able to provide verbal informed consent.

Payer/health insurance provider inclusion criteria:

* Employed at an organization or agency that provides funding for medical services for HIV-infected individuals for at least 6 months.
* Able to provide verbal informed consent.

Exclusion Criteria:

* Unable to provide verbal informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3838 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Fiellin, MD, Principal Investigator — Yale University; Jennifer Edelmen, MD, Study Director — Yale University
Locations (4):
- United States (4):
  - Hartford Hospital's HIV Clinic, Hartford, Connecticut
  - Haelen Center at Yale New Haven Hospital, New Haven, Connecticut
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Immunology Center at Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edelman EJ, Dziura J, Esserman D, Porter E, Becker WC, Chan PA, Cornman DH, Rebick G, Yager J, Morford K, Muvvala SB, Fiellin DA. Working with HIV clinics to adopt addiction treatment using implementation facilitation (WHAT-IF?): Rationale and design for a hybrid type 3 effectiveness-implementation study. Contemp Clin Trials. 2020 Nov;98:106156. doi: 10.1016/j.cct.2020.106156. Epub 2020 Sep 23. PMID 32976995
- [Result] Edelman EJ, Gan G, Dziura J, Esserman D, Morford KL, Porter E, Chan PA, Cornman DH, Oldfield BJ, Yager JE, Muvvala SB, Fiellin DA. Readiness to Provide Medications for Addiction Treatment in HIV Clinics: A Multisite Mixed-Methods Formative Evaluation. J Acquir Immune Defic Syndr. 2021 Jul 1;87(3):959-970. doi: 10.1097/QAI.0000000000002666. PMID 33675619
- [Result] Morford KL, Muvvala SB, Chan PA, Cornman DH, Doernberg M, Porter E, Virata M, Yager JE, Fiellin DA, Edelman EJ. Patients' perspectives of medications for addiction treatment in HIV clinics: A qualitative study. J Subst Abuse Treat. 2022 Aug;139:108767. doi: 10.1016/j.jsat.2022.108767. Epub 2022 Mar 18. PMID 35341613
- [Result] Edelman EJ, Gan G, Dziura J, Esserman D, Porter E, Becker WC, Chan PA, Cornman DH, Helfrich CD, Reynolds J, Yager JE, Morford KL, Muvvala SB, Fiellin DA. Effect of Implementation Facilitation to Promote Adoption of Medications for Addiction Treatment in US HIV Clinics: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2236904. doi: 10.1001/jamanetworkopen.2022.36904. PMID 36251291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At each of the 6 month assessment stages, the numbers fluctuate based on the number of patients identified in the electronic health record (EHR) and the number of clinicians and staff that completed each survey. The numbers at each stage are part of a sliding cohort where direct follow up with patients and clinicians longitudinally is not part of the design. Assessment of patients using EHR began 6 months prior to the assessment of clinicians and staff using surveys.
Units Other Than Participants: Clinics
Groups:
- Patient Characteristics: Patients from 4 clinics at each phase in the implementation facilitation design.
- Clinician/Staff Characteristics: Clinician/staff participants from 4 clinics at each phase phase in the implementation facilitation design.
Period: Overall Study
Arm/Group | Patient Characteristics | Clinician/Staff Characteristics
Started (Control Stage) | 3517; 4 Clinics (These are patients assessed through electronic health records and the number can fluctuate at each stage. These patient 'started' total numbers come from the control period prior to stage 1.) | 70; 4 Clinics (These are clinicians and staff assessed through surveys and the number can fluctuate at each period. These individuals 'started' totals comes from when they were assessed at the beginning of the first period in the study.)
Control Period | 4259; 4 Clinics (These are patients assessed through electronic health records and the number can fluctuate at each period.) | 69; 4 Clinics (These are clinicians and staff assessed through surveys and the number can fluctuate at each stage.)
Intervention Period | 3780; 4 Clinics (These are patients assessed through electronic health records and the number can fluctuate at each period.) | 59; 4 Clinics (These are clinicians and staff assessed through surveys and the number can fluctuate at each period.)
Evaluation Period | 3786; 4 Clinics (These are patients assessed through electronic health records and the number can fluctuate at each period.) | 58; 3 Clinics (These are clinicians and staff assessed through surveys and the number can fluctuate at each period. 1 site had an issue with provider follow up at this during this period.)
Maintenance Period | 4036; 4 Clinics (These are patients assessed through electronic health records and the number can fluctuate at each stage.) | 88; 4 Clinics (These are clinicians and staff assessed through surveys and the number can fluctuate at each period.)
Completed | 3514; 4 Clinics (These are patients assessed through electronic health records and the number can fluctuate at each period.) | 62; 4 Clinics (These are the clinicians and staff that were assessed through surveys during the final stage.)
Not Completed | 3; 0 Clinics | 8; 0 Clinics

BASELINE CHARACTERISTICS:
Population: These are counts of the participants (patients and clinician/staff) that were assessed at the end of the control stage (stage 1 in the participant flow).
Units Other Than Participants: Clinics
Groups:
- Patient Characteristics: Presented are the characteristics of patients across 4 clinics in the control (baseline) phase in the implementation facilitation design.
- Clinician/Staff Characteristics: Presented are the characteristics of clinician/staff participants across 4 clinics in the control (baseline) phase in the implementation facilitation design.
- Total: Total of all reporting groups
Arm/Group | Patient Characteristics | Clinician/Staff Characteristics | Total
Number analyzed (Participants) | 3647 | 70 | 3717
Number analyzed (Clinics) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12) | 58 (41) | NA (NA) — These are separate populations.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1407 | 51 | 1458
  Male | 2240 | 19 | 2259
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 781 | 12 | 793
  Not Hispanic or Latino | 2859 | 52 | 2911
  Unknown or Not Reported | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 19 | 6 | 25
  Race: Black | 1814 | 10 | 1824
  Race: White | 1118 | 45 | 1163
  Race: Other | 689 | 8 | 697
  Race: Missing | 7 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3647 | 70 | 3717
Public insurance [Count of Participants; unit: Participants] — Population: Patient Specific Measure
  Participants
    number analyzed (Participants) | 3647 | 0 | 3647
    Yes | 1725 |  | 1725
    No | 740 |  | 740
    Missing | 1182 |  | 1182
Self-Pay [Count of Participants; unit: Participants] — Patient Specific Measure: Self Paying Patient Population: Patient Specific Measure
  Participants
    number analyzed (Participants) | 3647 | 0 | 3647
    Yes | 21 |  | 21
    No | 2444 |  | 2444
    Missing | 1182 |  | 1182
Private or commercial insurance [Count of Participants; unit: Participants] — Patient Specific Measure: Insurance Type Population: Patient Specific Measure
  Participants
    number analyzed (Participants) | 3647 | 0 | 3647
    Yes | 985 |  | 985
    No | 1480 |  | 1480
    Missing | 1182 |  | 1182
Completed Visits at Baseline [Median (Full Range); unit: Clinic Visits] — Population: Patient Specific Measure
  Clinic Visits
    number analyzed (Participants) | 3647 | 0 | 3647
    (all) | 2 [0 to 17] |  | 2 [0 to 17]
Prescribed Antiretroviral Therapy [Count of Participants; unit: Participants] — Patients prescribed antiretroviral therapy at baseline. Population: Patient Specific Measure
  Participants
    number analyzed (Participants) | 3647 | 0 | 3647
    Yes | 3430 |  | 3430
    No | 217 |  | 217
Detectable HIV viral load (>200 copies/mL) [Count of Participants; unit: Participants] — Patients with detectable HIV viral load (>200 copies/mL). Population: Patient Specific Measure
  Participants
    number analyzed (Participants) | 3647 | 0 | 3647
    Yes | 325 |  | 325
    No | 2774 |  | 2774
    Missing | 548 |  | 548
Hepatitis C virus infection [Count of Participants; unit: Participants] — Patients with hepatitis C virus infection. Population: Patient Specific Measure
  Participants
    number analyzed (Participants) | 3647 | 0 | 3647
    Yes | 522 |  | 522
    No | 3072 |  | 3072
    Missing | 53 |  | 53
CD4 cell count categorized (cells/μL) [Count of Participants; unit: Participants] — Patients CD4 cell count (cells/μL) Population: Patient Specific Measure
  Participants
    number analyzed (Participants) | 3647 | 0 | 3647
    <50 | 31 |  | 31
    50-99 | 42 |  | 42
    100-199 | 154 |  | 154
    200-349 | 336 |  | 336
    350-499 | 480 |  | 480
    >500 | 1697 |  | 1697
    Missing | 907 |  | 907
Clinician (physicians, physician assistant, nurse practitioner) [Count of Participants; unit: Participants] — Clinician (physicians, physician assistant, nurse practitioner) yes or no Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    Yes |  | 34 | 34
    No |  | 36 | 36
Time working at clinic [Mean (Standard Deviation); unit: years] — Population: Clinician and Staff Participant Specific Measure
  years
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 7 (8) | 7 (8)
Time per week spent working at HIV clinic [Median (Full Range); unit: hours] — Population: Clinician and Staff Participant Specific Measure
  hours
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 31 [3 to 55] | 31 [3 to 55]
Ever prescribed medications to treat tobacco use disorder [Count of Participants; unit: Participants] — Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 32 | 32
Ever provided counseling to treat tobacco use disorder [Count of Participants; unit: Participants] — Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 34 | 34
Ever prescribed medications to treat unhealthy alcohol use [Count of Participants; unit: Participants] — Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 14 | 14
Ever provided counseling to treat unhealthy alcohol use [Count of Participants; unit: Participants] — Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 34 | 34
Ever provided counseling to treat opioid use disorder [Count of Participants; unit: Participants] — Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 32 | 32
Hold a waiver that allows buprenorphine (eg, Suboxone) prescribing [Count of Participants; unit: Participants] — Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 11 | 11
Ever prescribed oral or injectable (eg, Vivitrol) naltrexone to treat opioid use disorder [Count of Participants; unit: Participants] — Population: Clinician and Staff Participant Specific Measure
  Participants
    number analyzed (Participants) | 0 | 70 | 70
    (all) |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Provision of Addiction Treatments
Description: Study team will use the electronic health record (EHR) to identify prescriptions for each of the target medications in the surveillance period. Study team will use CPT codes to determine whether specific counseling therapies were provided. Patients diagnosed with Opioid Use Disorder and/or Alcohol Use Disorder and/or Tobacco Use Disorder were identified and then assessed in the EHR to determine if medication assisted therapy was provided by a provider during the 6 month Intervention period.
Time Frame: Baseline, 6 months
Population: Unduplicate count of participants from control stage to intervention stage.
Measure: Count of Participants; unit: Participants
Groups:
- Opioid Use Disorder Patients: Patients diagnosed with Opioid Use Disorder (OUD).
- Alcohol Use Disorder Patients: Patients diagnosed with Alcohol Use Disorder (AUD).
- Tobacco Use Disorder: Patients diagnosed with Tobacco Use Disorder
Arm/Group | Opioid Use Disorder Patients | Alcohol Use Disorder Patients | Tobacco Use Disorder
Number analyzed (Participants) | 277 | 296 | 955
Participants
  Control (Baseline): number analyzed (Participants) | 243 | 251 | 810
  Control (Baseline) | 66 | 20 | 268
  Intervention (6 months): number analyzed (Participants) | 117 | 122 | 444
  Intervention (6 months) | 33 | 15 | 183
Statistical Analysis 1: Comparison: Opioid Use Disorder Patients; Test type: Superiority; p = 0.55, Generalized Estimating Equation; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.82 to 1.45]
Statistical Analysis 2: Comparison: Alcohol Use Disorder Patients; Test type: Superiority; p = 0.09, Generalized Estimating Equation; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.92 to 3.37]
Statistical Analysis 3: Comparison: Tobacco Use Disorder; Test type: Superiority; p = 0.001, Generalized Estimating Equation; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.14 to 1.71]

2. Primary Outcome: Change in Provision of Addiction Treatments
Description: Study team will use the electronic medical record to identify prescriptions for each of the target medications in the surveillance period. Study team will use CPT codes to determine whether specific counseling therapies were provided. Patients diagnosed with Opioid Use Disorder and/or Alcohol Use Disorder and/or Tobacco Use Disorder were identified and then assessed in the EHR to determine if medication assisted therapy was provided by a provider during the 12 month Evaluation period.
Time Frame: Baseline, 12 months
Population: Unique patients assessed across the two time points by disorder type.
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Use Disorder Patients | Alcohol Use Disorder Patients | Tobacco Use Disorder
Number analyzed (Participants) | 299 | 293 | 993
Participants
  Control (Baseline): number analyzed (Participants) | 243 | 251 | 810
  Control (Baseline) | 66 | 20 | 268
  Evaluation (12 months): number analyzed (Participants) | 135 | 112 | 477
  Evaluation (12 months) | 38 | 15 | 190
Statistical Analysis 1: Comparison: Opioid Use Disorder Patients; Test type: Superiority; p = 0.59, Generalized Estimating Equation; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.81 to 1.45]
Statistical Analysis 2: Comparison: Alcohol Use Disorder Patients; Test type: Superiority; p = 0.11, Generalized Estimating Equation; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.88 to 3.55]
Statistical Analysis 3: Comparison: Tobacco Use Disorder; Test type: Superiority; p = 0.005, Generalized Estimating Equation; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.09 to 1.66]

3. Secondary Outcome: Antiretroviral Therapy (ART) Receipt
Description: ART receipt will be defined as at least 180 days of three concurrent antiretroviral agents in the 6-month interval based on prescriptions in the electronic medical record.
Time Frame: 6 months
Population: All those included in the multiple control and intervention phases across sites.
Measure: Count of Participants; unit: Participants
Groups:
- Control Period: Patients monitored during the control period.
- Intervention Period: Patients monitored during the intervention period.
Arm/Group | Control Period | Intervention Period
Number analyzed (Participants) | 4259 | 3780
Participants | 4106 | 3547

4. Secondary Outcome: Antiretroviral Therapy (ART) Receipt
Description: as for outcome 3
Time Frame: 12 months
Population: All patients monitored across all (multiple) control and evaluation periods.
Measure: Count of Participants; unit: Participants
Groups:
- Evaluation Period: Patients monitored during the evaluation period.
Arm/Group | Control Period | Evaluation Period
Number analyzed (Participants) | 4259 | 3786
Participants | 4106 | 3508

5. Secondary Outcome: Viral Suppression
Description: Viral suppression, will be defined as HIV RNA <200 copies/mL at last test closest to the time of data extraction, consistent with Department of Health and Human Services (DHHS) guidelines. Although current limits of detection are lower, this cutoff allows for low-level "blips" that have no clinical significance.
Time Frame: 6 months
Population: All patients monitored across all control (multiple) and intervention periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Period | Intervention Period
Number analyzed (Participants) | 4085 | 3165
Participants | 3849 | 2880

6. Secondary Outcome: Viral Suppression
Description: as for outcome 5
Time Frame: 12 months
Population: All patients monitored across all control (multiple) and evaluation periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Period | Evaluation Period
Number analyzed (Participants) | 4085 | 3138
Participants | 3849 | 2830

7. Secondary Outcome: VACS Index
Description: The Veterans Aging Cohort Study Index (VACS Index) creates a score by summing pre-assigned points for age, routinely monitored indicators of HIV disease (CD4 count and HIV-1 RNA), and general indicators of organ system injury including hemoglobin, platelets, aspartate and alanine transaminase (AST and ALT), creatinine, and viral hepatitis C infection (HCV). This score is weighted to indicate increasing risk of all-cause mortality with increasing score. The score can be used to estimate risk of all-cause mortality using a conversion factor. The VACS Index will be evaluated based on most recent values at the time of data extraction. VACS Index score will be treated as a continuous variable. VACS Index: minimum value: 0; maximum value: 164- a higher score means a worse outcome.
Time Frame: 6 months
Population: Unduplicated count of survey respondents at each administration.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Control Period: Providers surveyed during the control period.
- Intervention Period: Providers surveyed during the intervention period.
Arm/Group | Control Period | Intervention Period
Number analyzed (Participants) | 69 | 59
units on a scale | 23.53 [22.94 to 24.12] | 24.54 [23.76 to 25.32]

8. Secondary Outcome: VACS Index
Description: as for outcome 7
Time Frame: 12 months
Population: Unduplicated count of survey respondents at each administration.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Evaluation Period: Providers surveyed during the evaluation period.
Arm/Group | Control Period | Evaluation Period
Number analyzed (Participants) | 69 | 58
units on a scale | 23.53 [22.94 to 24.12] | 25.12 [24.31 to 25.94]

9. Secondary Outcome: Retention in HIV Care
Description: Retention in HIV care, per DHHS guidelines uses a 24-month measurement period. It is defined as at least one HIV medical care visit in each 6-month period, with a minimum of 60 days between the first medical visit in the prior 6-month period and the last medical visit in the subsequent 6-month period. This measure has good agreement with the Institute of Medicine indicator for retention in care and is an independent predictor of mortality. We will evaluate whether patients have had at least 1 visit in the 6-month period prior to time of data extraction.
Time Frame: 6 months
Population: Patients identified at the control period to follow up with at the end of the intervention period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Period
Number analyzed (Participants) | 4259
Participants | 3567

10. Secondary Outcome: Retention in HIV Care
Description: as for outcome 9
Time Frame: 12 months
Population: Patients identified at the control period to follow up with at the end of the evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluation Period
Number analyzed (Participants) | 4259
Participants | 3450

11. Secondary Outcome: Organizational Readiness
Description: Investigators will use the ORCA to measure factors impacting the provision of addiction treatments. This 15-minute survey is based on the PARiHS framework and asks the respondent to rate local factors related to evidence, context and facilitation on a 5-point Likert scale from strongly disagree to strongly agree. Facilitation questions will be omitted from the pre-implementation assessment since this part of the intervention and will not have taken place. The score has a range from 1 to 5 where a higher score indicates higher readiness.
Time Frame: 6 months
Population: Unduplicated count of survey respondents for the intervention period.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Opioid Use Disorder: Providers' ORCA rating for patients diagnosed with Opioid Use Disorder (OUD).
- Alcohol Use Disorder: Providers' ORCA rating for patients diagnosed with Alcohol Use Disorder (AUD).
- Tobacco Use Disorder: Providers' ORCA rating for patients diagnosed with Tobacco Use Disorder
Arm/Group | Opioid Use Disorder | Alcohol Use Disorder | Tobacco Use Disorder
Number analyzed (Participants) | 59 | 59 | 59
units on a scale | 4.46 [4.25 to 4.67] | 4.14 [3.91 to 4.37] | 4.31 [4.09 to 4.52]

12. Secondary Outcome: Organizational Readiness
Description: as for outcome 11
Time Frame: 12 months
Population: Unduplicated count of survey respondents for the maintenance period.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Opioid Use Disorder | Alcohol Use Disorder | Tobacco Use Disorder
Number analyzed (Participants) | 58 | 58 | 58
units on a scale | 4.37 [4.18 to 4.56] | 4.05 [3.86 to 4.24] | 4.13 [3.89 to 4.36]

13. Secondary Outcome: Provider Readiness
Description: Investigators will use change rulers, among appropriate providers, for each of the medications and counseling to assess readiness to provide each medication and counseling intervention. The change rulers will independently assess, on a 0-10 scale each provider's: 1) confidence to prescribe/provide the intervention, 2) readiness to prescribe/provide the intervention and 3) commitment to prescribe/provide the intervention. Presented is the score that indicates readiness to prescribe medication. The score has a range from 1 to 10 where a higher score indicates increased readiness.
Time Frame: 6 months
Population: Unduplicated count of survey respondents for the intervention period.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Opioid Use Disorder: Providers' readiness rating for patients diagnosed with Opioid Use Disorder (OUD).
- Alcohol Use Disorder: Providers' readiness rating for patients diagnosed with Alcohol Use Disorder (AUD).
- Tobacco Use Disorder: Providers' readiness rating for patients diagnosed with Tobacco Use Disorder
Arm/Group | Opioid Use Disorder | Alcohol Use Disorder | Tobacco Use Disorder
Number analyzed (Participants) | 59 | 59 | 59
units on a scale | 6.75 [5.93 to 7.57] | 6.22 [5.41 to 7.03] | 7.24 [6.49 to 8.00]

14. Secondary Outcome: Provider Readiness:
Description: Investigators will use change rulers, among appropriate providers, for each of the medications and counseling to assess readiness to provide each medication and counseling intervention.185 The change rulers will independently assess, on a 0-10 scale each provider's: 1) confidence to prescribe/provide the intervention, 2) readiness to prescribe/provide the intervention and 3) commitment to prescribe/provide the intervention. Presented is the score that indicates readiness to prescribe medication. The score has a range from 1 to 10 where a higher score indicates increased readiness.
Time Frame: 12 months
Population: Unduplicated count of survey respondents for the maintenance period.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Opioid Use Disorder | Alcohol Use Disorder | Tobacco Use Disorder
Number analyzed (Participants) | 58 | 58 | 58
units on a scale | 7.28 [6.47 to 8.10] | 7.16 [6.42 to 7.90] | 7.50 [6.69 to 8.32]

ADVERSE EVENTS:
Description: Adverse events were not collected as part of this study. The total 3759 is the largest number of patients assessed during the time period for the patient specific outcomes.
Groups:
- Patients: Patients from 4 clinics across all phases in the implementation facilitation design.
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT02907944/Prot_SAP_000.pdf